CLINICAL TRIAL: NCT00223210
Title: A Randomized, Double-Blind, Placebo-Controlled Add-On Trial of Quetiapine in Patients With Bipolar Disorder and Cocaine Dependence
Brief Title: An Add-On Trial of Quetiapine in Patients With Bipolar Disorder and Cocaine Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sherwood Brown, Dr. E. Sherwood Brown, PhD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRUSQUET 0397
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Bipolar Disorder; Cocaine Dependence
Keywords: bipolar disorder; cocaine dependence; quetiapine
MeSH Terms: conditions — Bipolar Disorder; Cocaine-Related Disorders | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quetiapine (Active Comparator)
  Interventions: Drug: Quetiapine
- Placebo (Placebo Comparator): Inactive ingredient matching the active medication in appearance
  Interventions: Drug: PLacebo

INTERVENTIONS:
Drug: Quetiapine — Active Quetiapine
  Other Names: Active Quetiapine
  Arms: Quetiapine
Drug: PLacebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if quetiapine add-on therapy is associated with a decrease in cocaine use and craving and a greater improvement in mood.

DETAILED DESCRIPTION:
One Hundred (100) outpatients with a diagnosis of bipolar I disorder and cocaine abuse/dependence, established by a structured clinical interview and confirmed by a psychiatrist, will participate. Eligible participants will be given a physical exam, including an eye exam with an ophthalmoscope to rule out serious medical illnesses and cataracts. Additionally, medical and psychiatric histories and baseline labs, including CBC and a liver panel will be obtained. Blood will be drawn for routine laboratory analyses including a complete blood count (CBC) and SMA-20 at baseline and exit. Women of childbearing potential will be given a urine pregnancy test. Baseline measures of psychiatric symptoms will be assessed with the Hamilton Rating Scale for Depression HRSD, Young Mania Rating Scale (YMRS), Inventory of Depression Symptomatology-Self-Report 30-item version (IDS-SR30), and the Psychobiology of Recovery in Depression III - Somatic Symptom Scale (PRD-III). Cocaine craving will be assessed with Cocaine Craving Questionnaire (CCQ). Drug use will be assessed by self-report, with the Addiction Severity Index (ASI) and a urine drug screen (UDS). Two UDSs are performed at baseline. Cocaine use in the past week (dollar amount spent/week and days used/week) will be assessed by patient self-report. Use of and craving for other substances (benzodiazepines, barbiturates, alcohol, opiates, phencyclidine, and cannabis) will also be assessed by self-report of dollar amount and days used in the past week, UDSs, and with 100-mm single item visual analog craving scales. Side effects will be assessed with the Abnormal Involuntary Movement Scale (AIMS), the Simpson-Angus Scale (SAS), and the Barnes Akathesia Rating Scale (BARS). Subjects will be randomized and be titrated up to 400 mg/day with additional flexible titration after that time to a maximum of 800 mg/day of Quetiapine or identical appearing placebo add-on therapy in a double- blind fashion for 12 weeks. At each weekly assessment subjects will be evaluated with the HRSD17, IDS-R30, YMRS, CCQ, and a UDS, and receive an upward titration of the study drug. The ASI will be repeated every four weeks. Further, participants will return one additional time each week for a UDS. At the end of the study an unblinded psychiatrist will provide standard open label treatment with Quetiapine until the participants can be transferred back to their usual treatment facility. Follow up and after care arrangements will be made for each participant near completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar Disorder, type I; Cocaine Dependence with use in the past 7 days; Currently taking a mood stabilizer; Meets criteria for a hypomanic or manic episode

Exclusion Criteria:

* Bipolar Disorder, type II, NOS; Cyclothymia; Other substance dependence; Diabetes; Initiated therapy in the past 2 weeks; History of cataracts or likely cataracts; Current active suicidal or homicidal ideation; Life threatening medical condition; Mental retardation, dementia or severe cognitive impairment; Pregnant or nursing womenon; antipsychotic within 7 days of beginning Quetiapine therapy or have initiated antidepressants or mood stabilizers or psychotherapy within the past two weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2005-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
A random regression analysis will be done with treatment group as the between-subjects factor, time as the within-subjects factor, and a group by time interaction. | Study Exit
Within-group differences between pre- and post- treatment of the study drug will be compared using Wilcoxon rank sum tests, if the sample is not normally distributed between-group differences will be compared using the Mann-Whitney test. | Study Exit
To identify response versus non-response, logistic regression, assuming linearity, will be used. | Study Exit
We will utilize the urine drug screen repeatedly and cocaine use/cravings as the primary outcome measure. | Study Exit
Changes from base line to exit for all patients finishing at-least one follow up of active Quetiapine therapy, will be calculated, using the last observation carried forward (LOCF). | Study Exit

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, MD, PhD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States